CLINICAL TRIAL: NCT06198127
Title: Effects of Core Stability Exercises With and Without Kinesio-taping on Trunk Control, Gait and Posture in Children With Cerebral Palsy
Brief Title: Effect of Core Stability Exercises With and Without Kinesio-Taping in CP Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0748
Record Dates: First submitted 2023-12-26; First posted 2024-01-10 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Spastic Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: The study will be randomized controlled trial used to determine the effect of core stability exercises with and without kinesio-taping in CP children. Subjects with CP meeting the pre-determined inclusion and exclusion criteria will be divided into two groups using non-probability sampling technique.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group; combination of core stability exercises and kinesio-taping (Experimental): combination of core stability exercises and kinesio-taping were used in experimental group
  Interventions: Other: combination of core stability exercises and kinesio-taping
- Control group; only core stability exercises (Active Comparator): only core stability exercises were given to control group
  Interventions: Other: Core stability exercises

INTERVENTIONS:
Other: combination of core stability exercises and kinesio-taping — the patient in the experimental group will receive the core stability exercises with kinesiology taping on trunk stabilizer muscles. the time of intervention was 30 minutes per day. The exercises such as Abdominal draw-in with a double knee to chest, Trunk twist while sitting on a medicine ball, Lying in a supine position on bed and rotating the trunk from side-to-side, Bridging exercises, the I-shaped elastic KT will apply to the four trunk muscles from their insertion to their origin: Kinesio-taping is used on global muscles such as Rectus abdominis, External obliques, Erector spinae, Quadratus lumborum. Kinesio-taping will 1 inch wide and apply on muscles for 1 to 2 days then remove for 24 hours then again apply a new one. The tension will be 10 to 15% and tape will apply on muscles which will be stretched by maintaining a posture.
  Arms: Experimental group; combination of core stability exercises and kinesio-taping
Other: Core stability exercises — After the baseline assessment, the patient in the control group will receive the core stability exercises with kinesio-taping on trunk stabilizer muscles. Time of rehabilitation will be 30 minutes per subject and four days per week. In first few minutes, the subject will be explained her/his task Subject will execute the exercises such as Abdominal draw-in with a double knee to chest 10- 15 times. Trunk twist while sitting on a medicine ball 10- 15 times. Lying in a supine position on bed and rotating the trunk from side-to-side 10- 15 times. Lying in a supine position on a mat and pulling upper and lower limbs upward 10- 15 times. Bridging exercises 10- 15 times, Deep Breathing and Wheelbarrow.
  Arms: Control group; only core stability exercises

SUMMARY:
Cerebral Palsy (CP) is a motor disorder caused by damage to the brain that affects posture, movement, and muscle control. It can lead to difficulties with trunk control, gait, and posture, which can impact daily activities and quality of life. Core stability exercises have been shown to improve trunk control, gait, and posture in children with CP by improving muscle activation patterns and enhancing postural stability. Kinesio-taping, on the other hand, is a therapeutic technique that involves the application of a stretchy tape to the skin to provide support, stability, and pain relief to the muscles and joints. It has been proposed that kinesio-taping may enhance the effects of exercises by providing additional support and proprioceptive feedback.

This will be randomized controlled trial study. Sampling technique will be non-probability convenience sampling. Computer randomization will be used to locate subjects in two groups. After that informed consent will be taken and patients will be included in the study based on the inclusion criteria. Study will be conducted in 22 CP children age 7-12 years, ability to stand and walk, ability to follow instructions and assess by assessment tools as GMFCS level II, GARS, TIS and PAS pre and post intervention. Study groups will be divided into 2 groups, Group A (study Group) and group B (control group) Group A: Experimental group; combination of core stability exercises and kinesio-taping Group B: control group; only core stability exercises. Data will be analyzed by using SPSS-25. Appropriate statistical test will be used after checking normality of data.

DETAILED DESCRIPTION:
Experimental Group:

After the baseline assessment, the patient in the experimental group will receive the core stability exercises with kinesio-taping on trunk stabilizer muscles. Time of rehabilitation will be 30 minutes per subject and four days per week. In first few minutes, the subject will be explained her/his task Subject will execute the exercises such as Abdominal draw-in with a double knee to chest 10- 15 times. Trunk twist while sitting on a medicine ball 10- 15 times. Lying in a supine position on bed and rotating the trunk from side-to-side 10- 15 times. Lying in a supine position on a mat and pulling upper and lower limbs upward 10- 15 times. Bridging exercises 10- 15 times. Deep Breathing and Wheelbarrow.(4) Kinesio-taping: The area to be taped will be cleaned with an alcohol swab, and the I-shaped elastic Kinesio-taping will apply to the four trunk muscles from their insertion to their origin: Kinesio-taping is used on global muscles such as Rectus abdominis, External obliques, Erector spinae, Quadratus lumborum. For the rectus abdominis (RA) muscle, the kinesio-taping will be applied from the xiphoid process and the fifth to seventh costal cartilages to near the pubic symphysis in the hooking position. For the external oblique (EO) muscle, the kinesio-taping will be applied from the inguinal region to the T12 spinous process in the side-lying position, and for the internal oblique (IO) muscle, the kinesio-taping will be applied from the xiphoid process to the anterior half of the crest of the ilium in the same position. For the erector spinae muscle, the kinesio-taping will be applied from the ipsilateral transverse process of T12 to the posterior sacrum iliac crest. Kinesio-taping will 1 inch wide and apply on muscles for 1 to 2 days then remove for 24 hours then again apply a new one. The tension will be 10 to 15% and tape will apply on muscles which will be stretched by maintaining a posture .

Control Group :

After the baseline assessment, the patient in the control group will receive the core stability exercises with kinesio-taping on trunk stabilizer muscles. Time of rehabilitation will be 30 minutes per subject and four days per week. In first few minutes, the subject will be explained her/his task Subject will execute the exercises such as Abdominal draw-in with a double knee to chest 10- 15 times. Trunk twist while sitting on a medicine ball 10- 15 times. Lying in a supine position on bed and rotating the trunk from side-to-side 10- 15 times. Lying in a supine position on a mat and pulling upper and lower limbs upward 10- 15 times. Bridging exercises 10- 15 times, Deep Breathing and Wheelbarrow .

ELIGIBILITY:
Inclusion Criteria:

* Aged 7-12 years participants
* Children with spastic CP.
* Have ability to keep balance in standing position and take steps without support according to GMFCS level ii.
* Have ability to follow commands of the examiner

Exclusion Criteria:

* allergy to kinesiology taping,
* Skin diseases such as eczema or psoriasis, congenital curve or due to (neuromuscular, rheumatologic, renal, cardiovascular, pulmonary, or vestibular diseases),
* patients with metabolic, infectious, traumatic conditions, psychological, psychiatric problems,
* subjects with any other disorders which lead to changes in spinal curves or any back disorders, such as spondylolysis, spondylolisthesis and lumbosacral transitional anomalies
* fixed contracture or deformities in the spine or extremities, visual or respiratory disorders

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Trunk control with the Trunk Impairment Scale | 6 weeks
  The Trunk Impairment Scale (TIS) measures static and dynamic seated trunk control in children with cerebral palsy (CP) who have postural control problems. TIS consists of 17 items in three subscales: static sitting balance, dynamic sitting balance, coordination with a total score range of 0 to 23 points.
Posture and Postural ability scale (PPAS) | 6 weeks
  The Posture and Postural Ability Scale is a 7-point ordinal scale for the assessment of postural ability. There are six items for assessment of quality of posture in the frontal plane and another six items in the sagittal plane.
Gait abnormality rating scale (GARS) | 6 weeks
  Gait Abnormality Rating Scale (GARS) is a videotape-based analysis of 16 facets of human gait. The Gait Abnormality Rating Scale was designed to observe the gait pattern of older adults with increased fall risk. This scale examines the interaction of the trunk, and upper and lower limb movements during walking. It also includes items that reflect the walking speed and stride length, traditional temporospatial gait parameters, The GARS scale puts more emphasis on assessing overall functional performance. For the elderly, this scale sensitively indicates their deficits during walking and is related to increased fall risk. the intra-rater and inter-rater reliabilities of the total GARS score is 0.708 and 0.875 which is acceptable.

CONTACTS AND LOCATIONS:
Overall Officials: Alina Amjad, MS*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kamel MI, Sayed Elawh Moubarak EE, El-Nassag BA, El-Hakim A-M, Abdulrahman RS. Effects of core stabilization exercise and kinesio taping on pain, Cobb angle and endurance of trunk muscles in children and adolescents with idiopathic scoliosis. Curr Pediatr Res [Internet]. 2022;26(3):1289-1297. Available from: https://www.cochranelibrary.com/central/doi/10.1002/central/CN-02474713/full
- [Background] Lee H, Lim H. Effects of Double-Taped Kinesio Taping on Pain and Functional Performance due to Muscle Fatigue in Young Males: A Randomized Controlled Trial. Int J Environ Res Public Health. 2020 Mar 31;17(7):2364. doi: 10.3390/ijerph17072364. PMID 32244424